CLINICAL TRIAL: NCT00427674
Title: Phase I Evaluation of (123-I)MZINT as a Brain SPECT Tracer of Serotonin Transporters in Healthy Human Subjects
Brief Title: Assessment of the Biodistribution and Safety of 123-I MZINT in Healthy Subjects and Parkinson Disease Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Scan results to date did not show reason to continue with study
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: Molecular NeuroImaging (Other)
Responsible Party: John Seibyl, MD, MNI
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: _mZINT_001/002
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2010-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Imaging
MeSH Terms: conditions — Parkinson Disease | interventions — Iodine-123

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- injection of 5 mCi of 123-I mZINT (Experimental)
  Interventions: Drug: [123I] mZINT injection and serial dynamic SPECT imaging

INTERVENTIONS:
Drug: [123I] mZINT injection and serial dynamic SPECT imaging — Following bolus intravenous injection of 5 mCi of 123-I mZINT over 15 seconds, serial dynamic SPECT brain acquisitions will be obtained to evaluate the regional brain uptake and washout of activity. Venous blood measures will be obtained with each acquisition and characterization of 123-I mZINT and metabolites will be assessed. Safety assessments will include vital signs, serum chemistries, CBC, urinalysis, and EKG.

SUMMARY:
The overall plan of this project is to evaluate [123I] mZINT as a tool to assess SERT density in humans. This protocol will be completed in three parts. In Part A serial dynamic SPECT will be acquired after injection of [123I] mZINT in healthy controls to assess regional brain uptake in human subjects. If Part A demonstrates robust brain region specific uptake, then Part B - additional studies in healthy subjects to assess biodistribution, and Part C - studies in PD subjects to compare regional uptake to healthy controls, will be completed.

DETAILED DESCRIPTION:
All study procedures will be conducted at the Institute for Neurodegenerative Disorders (IND) and Molecular NeuroImaging (MNI) in New Haven, CT. Approximately 10 (6 -Part A and 4 - Part B) healthy subjects and 10 PD subjects will be recruited from the IND databases, patient spouses, and the community to participate in this protocol. The study doctor will discuss the study procedures and evaluate the subject for eligibility. All subjects will undergo written informed consent and a screening evaluation including baseline clinical laboratory testing, and a baseline physical and neurological evaluation.

Following bolus intravenous injection of 5 mCi of 123-I mZINT over 15 seconds, serial dynamic SPECT brain acquisitions will be obtained to evaluate the regional brain uptake and washout of activity. Venous blood measures will be obtained with each acquisition and characterization of 123-I mZINT and metabolites will be assessed. Safety assessments will include vital signs, serum chemistries, CBC, urinalysis, and EKG.

Vital signs will be assessed at pre-injection baseline and 15, 30, 60, and 90 minutes following the infusion of 123-I mZINT. An EKG will be obtained at baseline and at 20 and 40 min post 123-I mZINT injection. Adverse events will be assessed when vital signs are obtained. Clinical laboratory tests performed at baseline and after each injection including the following: serum chemistry battery, complete blood count with differential, and urinalysis.

ELIGIBILITY:
Inclusion Criteria:

Health Control:

* The subject is aged 18-70.
* Written informed consent is obtained.
* The participant has no clinically significant clinical laboratory value and/or clinically significant unstable medical, neurological or psychiatric illness.
* For females, non-child bearing potential or negative urine pregnancy test on day of [123I] mZINT injection.
* Willingness to comply with the study protocol

Parkinson disease:

* The subject is aged 18-70.
* Participants have a clinical diagnosis (at least two of the three cardinal symptoms: resting tremor, rigidity, bradykinesia) of idiopathic Parkinson's disease.
* Hoehn and Yahr stages < 3.
* Written informed consent is obtained.
* The participant has no clinically significant clinical laboratory value and/or clinically significant unstable medical, neurological or psychiatric illness.
* For females, non-child bearing potential or negative urine pregnancy test on day of [123I] mZINT injection.

Willingness to comply with the study protocol

Exclusion Criteria:

All Subjects will be excluded from participation for the following reasons:

* The subject has a clinically significant clinical laboratory values abnormality, and/or medical or psychiatric illness.
* The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery).
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Use of all prescription drugs or non-prescriptions drugs that may effect serotonin such as antidepressants including sertraline, fluoxetine, fluvoxamine, venlafaxine.
* The participant has a history of alcohol, narcotic, or any other drug abuse as defined by the Diagnostic and Statistical Manual of the American Psychiatric Association, 4th Edition (DSM IV) {American Psychiatric Association, 1994 #2} within the past 2 years.
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-01; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Measurement of 123-mZINT brain uptake and distribution | 1 yr
pharmacokinetics of brain uptake and washout | 1 year
measurement of biodistribution and radiation absorbed dose of 123-I MZINT in the brain SERT | 1 yr
Evaluation for reduction in midbrain and/or striatal SERT density using 123-I MZINT. | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: John P Seibyl, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States